CLINICAL TRIAL: NCT03375749
Title: StandUP UBC: Impact of a Low-cost Standing Desk on Reducing Workplace Sitting
Brief Title: StandUP UBC: Reducing Workplace Sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Guy Faulkner, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H17-02776
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Sedentary Lifestyle
Keywords: sitting
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing Desk Intervention (Experimental): Each participant allocated to the experimental group will receive a low-cost, cardboard, fixed-height standing desk converter (https://oristand.co/) that will be placed in their regular office environment, along with their usual sitting desk. The participants will be instructed on how to use the fixed-height standing desk converter (herein referred to as standing desk) as a way to break up sitting time every 30 minutes. In addition, each participant will be provided with information about the health benefits of breaking up sitting time.
  Interventions: Behavioral: Standing desk intervention
- Waitlist Control (Other): Control group participants will not encounter any changes to their regular office environment. They will be provided with the standing desk and behaviour change strategies 6-months post-intervention.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Standing desk intervention — Standing desk converter
  Arms: Standing Desk Intervention
Behavioral: Waitlist control — Control
  Arms: Waitlist Control

SUMMARY:
Research indicates that sedentary behaviours, such as prolonged sitting, have negative health consequences and increases risk for disease. Unfortunately, many office-workers spend a high proportion of their workday sitting, often in prolonged unbroken bouts. Recent interventions have provided active workstations (e.g., sit-stand desks) to reduce employee sitting. However, cost prohibits provision of these desks in work environments. There is a need for low-cost solutions to reduce sitting at work. The purpose of this study is to determine whether provision of a low-cost standing desk reduces workplace sitting, and results in improvements in work engagement and fatigue, compared to usual practice.

DETAILED DESCRIPTION:
Study objectives: This study aims to provide a cost-effective solution to reducing sitting time during the workday, through provision of (1) low-cost cardboard standing desks ($20), and (2) simple behaviour change strategies (e.g., instruction on how to break up sitting time and information on the health consequences of doing so).

Background: Sedentary behaviour, defined as 'any waking behaviour characterised by an energy expenditure ≤1.5 metabolic equivalents while in a sitting, reclining, or lying posture', is a risk factor for poor health, independent of moderate-to-vigorous physical activity (MVPA). High levels of sedentary behaviour and excessive bouts of prolonged sitting is associated with increased risk for developing type 2 diabetes, cardiovascular disease and some cancers.

Sedentary behaviours are prevalent among Canadian adults, who often spend a large proportion of their waking hours sitting (e.g., work, commuting, watching TV), and office workers have been identified as one of the most sedentary occupational groups. Sedentary behaviour can be reduced by replacing sitting time with standing or light ambulation. In order to do so, it is vital to create an environment that makes sitting less likely and standing/moving easier. There is some evidence that introduction of sit-stand desks can reduce occupational sitting time within office environments ; however, there are cost barriers to the provision of these desks in work environments and few randomized control trials have demonstrated the long-term compliance and effectiveness of these desks on health- (e.g., weight, waist circumference, blood-derived biomarkers, musculoskeletal symptoms, fatigue) and work-related (e.g., work performance/productivity) outcomes. These are important factors that need to be considered and studied in further detail to quantify the benefit of sit-stand workstations.

Therefore, the purpose of this study is to evaluate the long-term effectiveness of a low-cost intervention aimed at reducing workplace sitting time in office workers.

Primary objectives:

• To evaluate the effectiveness of the intervention at reducing daily occupational sitting time over 6 months.

Secondary objectives:

• To explore whether the intervention results in improvements in work engagement and productivity, and occupational fatigue.

Methods/Design: The intervention will be delivered and evaluated over a 6-month period. This study is a two-arm randomized waitlist-controlled trial with one intervention group and one control group. After eligibility assessment, individuals will be randomly allocated to either the intervention or the control arm. The experimental group participants will receive a low-cost cardboard standing desk converter in their regular office environment and behaviour change strategies to break up sitting time, while the control group participants will not encounter any change to their regular work environments or be provided with any behaviour change strategies.

Intervention for experimental group:

Each participant allocated to the experimental group will receive a low-cost, cardboard, fixed-height standing desk converter (https://oristand.co/) that will be placed in their regular office environment, along with their usual sitting desk. The participants will be instructed on how to use the fixed-height standing desk converter (herein referred to as standing desk) as a way to break up sitting time every 30 minutes. In addition, each participant will be provided with information about the health benefits of breaking up sitting time.

Waitlist Control group:

Control group participants will not encounter any changes to their regular office environment. They will be provided with the standing desk and behaviour change strategies 6-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* (1) individuals who are desk-based (>75% of seated working hours),
* (2) work at least three days a week using the same desk,
* (3) aged 18-64 years, and
* (4) have the capability of standing.

Exclusion Criteria:

* (1) individuals who are not predominantly desk-based (<75% seated working hours),
* (2) work less than three days a week in the same office, or will not be working for the full duration of the study (i.e., retirement, term-time only, maternity/extended leave),
* (3) self-report having severe musculoskeletal conditions which restrict them from standing,
* (4) already use a standing desk.
* (5) unable to read or understand English or provide full informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Reduction in sitting time | Baseline, 3 months and 6 months
  Daily minutes sitting time measured with an activPAL3 micro activity monitor
Reduced number of prolonged sitting bouts (>30 min) | Baseline, 3 months and 6 months
  Number of daily bouts of sitting (>30 mins) measured with an activPAL3 micro activity monitor

SECONDARY OUTCOMES:
Work engagement | Baseline, 3 months and 6 months
  Utrecht Work Engagement Scale (UWES). Work engagement will be measured using the Utrecht Work Engagement Scale (UWES), a 7-point likert scale ("never" [0]to "always" [6]). There are three sub-scales: vigour, dedication, and absorption. The mean scale score of the three UWES subscales is computed by adding the 3 scores on each particular scale and dividing the sum by the number of items of the subscale involved. A similar procedure is followed for the total score. Hence, the UWES yields three subscale scores and/or a total score that range between 0 and 6. Higher values reflect better outcomes.
Occupational fatigue | Baseline, 3 months and 6 months
  Need for Recovery (NFR) scale. Occupational fatigue will be measured using the 11-item Need for Recovery (NFR) scale. Indicators of fatigue assessed on the NFR scale include a lack of concentration and reduced motivation for activities at the end of the day. Participants are given dichotomous response options (yes/no) to answer whether or not they experience each indicator. The total number of indicators present for each individual is converted into a scale score which ranges from 0 to 100, where higher scores show a greater need for recovery and thereby greater short-term work-related fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Faulkner, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tremblay MS, Aubert S, Barnes JD, Saunders TJ, Carson V, Latimer-Cheung AE, Chastin SFM, Altenburg TM, Chinapaw MJM; SBRN Terminology Consensus Project Participants. Sedentary Behavior Research Network (SBRN) - Terminology Consensus Project process and outcome. Int J Behav Nutr Phys Act. 2017 Jun 10;14(1):75. doi: 10.1186/s12966-017-0525-8. PMID 28599680
- [Background] Shrestha N, Kukkonen-Harjula KT, Verbeek JH, Ijaz S, Hermans V, Bhaumik S. Workplace interventions for reducing sitting at work. Cochrane Database Syst Rev. 2016 Mar 17;3(3):CD010912. doi: 10.1002/14651858.CD010912.pub3. PMID 26984326
- [Background] Neuhaus M, Eakin EG, Straker L, Owen N, Dunstan DW, Reid N, Healy GN. Reducing occupational sedentary time: a systematic review and meta-analysis of evidence on activity-permissive workstations. Obes Rev. 2014 Oct;15(10):822-38. doi: 10.1111/obr.12201. Epub 2014 Jul 11. PMID 25040784
- [Derived] Faulkner G, Weatherson KA, Duncan MJ, Wunderlich KB, Puterman E. Exploring Work-Time Affective States Through Ecological Momentary Assessment in an Office-Based Intervention to Reduce Occupational Sitting. J Phys Act Health. 2023 Apr 10;20(6):566-570. doi: 10.1123/jpah.2022-0495. Print 2023 Jun 1. PMID 37037458
- [Derived] Weatherson K, Yun L, Wunderlich K, Puterman E, Faulkner G. Application of an Ecological Momentary Assessment Protocol in a Workplace Intervention: Assessing Compliance, Criterion Validity, and Reactivity. J Phys Act Health. 2019 Nov 1;16(11):985-992. doi: 10.1123/jpah.2019-0152. Epub 2019 Sep 20. PMID 31541068
- [Derived] Weatherson KA, Wunderlich KB, Faulkner GE. Impact of a low-cost standing desk on reducing workplace sitting (StandUP UBC): A randomised controlled trial. Appl Ergon. 2020 Jan;82:102951. doi: 10.1016/j.apergo.2019.102951. Epub 2019 Sep 14. PMID 31526916